CLINICAL TRIAL: NCT06996899
Title: Establishing Utility of a Physical Health Improvement Intervention in a Regional Mental Health Impatient Service: a Multimethod Study
Brief Title: Physical Health Improvement Intervention for People Admitted to Mental Health Service
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charles Darwin University (Other)
Responsible Party: Principal Investigator, Nicole Norman, Principle Investigator (PhD Candidate), Registered Nurse, Charles Darwin University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H24039
Record Dates: First submitted 2024-12-13; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Physical Health; Mental Illnesses; Chronic Diseases
Keywords: Implementation Research; Health Improvement Profile
MeSH Terms: conditions — Mental Disorders; Chronic Disease | interventions — Potentially Inappropriate Medication List; Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: The one group is all adults admitted to the inpatient mental health service . The parallel group is the clinicians/staff working in the patient mental health service.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clinician/Staff users of the Health Improvement Profile (Experimental): Experimental: Staff intervention group Participants will receive education and training on how to conduct comprehensive physical assessments for the 27 health parameters on the Health Improvement Profile (HIP) and how to use these assessment finding to determine the recommended actions (behaviours changes) to develop an individualised profile for the admitted patient.
  Interventions: Other: Clinician Health Improvement Profile user training
- Experimental: Client receiving the Health Improvement Profile (Experimental): Experimental: Client intervention group Participants will have a comprehensive physical assessment conducted by a trained clinician (health professional in the mental health inpatient service. The assessments consist of 27 health parameters such as weight, Body Mass Index (BMI), blood pressure, blood glucose, cholesterol levels, and waist circumference, alongside questions on lifestyle factors like smoking, diet, and physical activity, as well as medication use and its side effects.
  Using the assessment data clients will participate in the development of an individualised Health Improvement Plan (HIP) utilising the recommended behaviour change actions.
  Interventions: Other: Health Improvement Profile (HIP)

INTERVENTIONS:
Other: Health Improvement Profile (HIP) — The Health Improvement Profile (HIP) is a comprehensive physical assessment conducted by a trained clinician which aims to link evidence based interventions for flagged abnormal health parameters. There are 27 health parameters assessed such as weight, Body Mass Index (BMI), blood pressure, blood glucose, cholesterol levels, and waist circumference, alongside questions on lifestyle factors like smoking, diet, and physical activity, as well as medication use and its side effects.
  Client participant will collaborate with their clinician in developing an individualised Health Improvement Profile which identifies suitable health behaviours interventions to improve physical health.
  Health behaviours may be associated with diet, exercise, sleep, hygiene (including oral care) and mindfulness.
  Other Names: Screening tool; motivational interviewing; behaviour change tool
  Arms: Experimental: Client receiving the Health Improvement Profile
Other: Clinician Health Improvement Profile user training — Clinician/staff participants will receive Health Improvement Profile user training on how to conduct the comprehensive physical assessments for 27 health parameters and how to link the evidence based actions to develop an individualised Health Improvement Profile for clients admitted to inpatient service. Training includes online videos simulating assessments and completing the Health Improvement Profile and face to face workshops.
  Arms: Clinician/Staff users of the Health Improvement Profile

SUMMARY:
This study aims to codesign and implement a physical health improvement behaviour change intervention for people being treated for a mental illness in a mental health inpatient unit of a regional hospital.

DETAILED DESCRIPTION:
People in regional areas with mental illness suffer high prevalence of preventable chronic health conditions. Multi-morbidity in people with mental illness contributes to a reduced life expectancy of up to 20 years. Many physical diseases are preventable and/or reversable if risk factors are identified early, and the right health promotion tools and interventions are provided. Addressing such a complex issue for people with mental illness requires an approach which is adaptable, has been co-designed with clinicians and consumers and is comprehensive to target individualised health behaviours.

This research uses the Health Improvement Profile (HIP) tool to help clinicians (e.g. nurses, doctors) to assess patients physical health and identify risk factors or early signs of chronic disease. Using the Health Improvement Profile (HIP) tool during admission the clinicians will work with clients to implement the most suitable health promotion tools to help improve physical health.

Using implementation research methodology and following the Consolidated Framework for Implementation Research (CFIR) the study is broken into the following 4 stages:

* Identify
* Adapt - codesign/adapt Health Improvement Profile (HIP) intervention and develop user training
* Implement - into clinical areas to assist developing personalised Health Improvement Profile (HIP)
* Evaluate - using both qualitative and quantitative data to determine feasibility of the Health Improvement Profile (HIP) and implementation in a regional health service

ELIGIBILITY:
Inclusion Criteria:

* This study is being carried out in an inpatient service therefore clinical staff must be registered by their professional governing body with a minimum of 6 months employment at the service or within the region to participate in stages 2 and 3. Graduate clinicians with less than 6 months working experience will be excluded from the study. Clinicians new to the region with less than 6 months working experience in location will be excluded from the study. Clinical roles within the facility include but not limited to:

  * Nurses (enrolled or registered)
  * Psychiatrists
  * Psychologists
  * Social Workers

Clients of the inpatient mental health service eligible to be included in the study must be:

* Over the age of 18 years
* Able to read, understand and speak English
* A current or previous user of the hospital's services
* A current or previous user of the inpatient services
* A carer of someone who is a current or previous user of the inpatient mental health service
* Able to provide consent
* Not an employee
* Not a health professional

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Health Improvement Profile | From admission (enrolment) to post discharge period of 3 months (12 weeks)
  Each Health Improvement Profile parameter has a column for recording the assessment result, followed by a column indicating the healthy 'green' range or indicating the unhealthy 'red' range (requiring action). The final column indicates the recommended action if the parameter falls into the 'red' range.
  Baseline assessment, (up to 27 assessment points for males and 26 assessment points for females) using the Health Improvement Profile (HIP) to identify the number of red flags, this is baseline assessment data which falls outside of normal healthy parameters.
  Baseline assessment will occur at pre intervention (at time of admission to the inpatient unit), during intervention use (at discharge from inpatient facility with a developed Health Improvement Profile) and post intervention (3months post discharge from inpatient facility) to determine physical health improvement against baseline assessment.
Feasibility: Time taken to recruit planned sample | Immediately after the inclusion of the last participant
  The time that was taken to recruit the planned sample size of participants
Feasibility: Retention | at the follow-up assessment 3 months post discharge from inpatient service
  Proportion of participants who completed the whole study by all participants who enrolled
Feasibility: Drop out rate | At the follow-up assessment 3 months post discharge from inpatient service
  Number of participants who dropped out , did not continue with health improvement profile after discharging from inpatient service
Reason for dropping out | immediately on drop out notification or at 3 month follow up
  Feedback from participant to identify reason for dropping out
Feasibility: Adherence | Immediately on completion of the post discharge period at 3 months (12 weeks)
  Proportion (percentage %) of recommended actions on the Health Improvement Profile (HIP) which the patient self reports as completing up to 3 months post discharge.
Participant feedback | Immediately after completion of the follow up period of 3 months (12 weeks)
  Participant qualitative feedback using open ended questions on satisfaction with the Health Improvement Profile. Analysed using standardised thematic analysis of the qualitative feedback.

SECONDARY OUTCOMES:
Clinician Confidence | At completion of training, at the project interim point (3 months) and at end of project.
  Participant qualitative feedback using open ended questions on confidence for clinicians undertaking the physical assessments and developing care plans
Client wellbeing | Immediately at completion of the follow up period (3 months)
  Participant qualitative feedback using open ended questions via interview or focus group, on self general overall self reported wellbeing physically and mentally (no quantitative scale to be used), this is qualitative feedback on client wellbeing participating in the HIP project.
Biometric measure: Body Mass Index (BMI) | At commencement (admission) to inpatient unit and after completion of follow up period 3 months (12 weeks)
  BMI (kg/m2) is calculated by dividing a person weight in kilograms by the square of their height in metres Outside of normal parameters (red flagged) Underweight <18.50 Overweight ≥25.00
Biometric measure: Waist circumference | At commencement (admission) to inpatient unit and after completion of follow up period at 3 months (12weeks)
  Measured in centimetres (cm) - measured by applying the tap measure midway between the top of the hip bone and bottom of ribs, in line with the belly button, wrap measuring tap around your waist.
  Outside of normal measure (red flagged) Female >80cm Male >94cm
Biometric measure: Pulse | At commencement (admission) to inpatient unit and after completion of follow up period at 3 months (12weeks)
  Beats per minute (BPM) Outside of normal parameters (red flagged) <60bpm/>100bpm
Biometric measure: Blood pressure | At commencement (admission) to inpatient unit and after completion of follow up period at 3 months (12weeks)
  Outside of normal parameters (red flagged) ≥140/90 millimeters of mercury (mm Hg)
Biometric measure: Temperature | At commencement (admission) to inpatient unit and after completion of follow up period at 3 months (12weeks)
  Outside of normal parameters (red flagged) <36°Celcius >37.5°Celcius
Biometric measure: Liver Function Test | At commencement (admission) to inpatient unit and after completion of follow up period at 3 months (12weeks)
  Outside of normal parameters (red flagged) Liver function test (LFTs) - components.
  • Alanine aminotransferase (ALT) IU/L;
Biometric measure: Liver Function Test | At commencement (admission) to inpatient unit and after completion of follow up period at 3 months (12weeks)
  Outside of normal parameters (red flagged) Liver function test (LFTs) - components.
  • Alkaline phosphatase (ALP) IU/L;
Biometric measure: Liver Function Test | At commencement (admission) to inpatient unit and after completion of follow up period at 3 months (12weeks)
  Outside of normal parameters (red flagged) Liver function test (LFTs) - components.
  • Gamma- glutamyl transferase (GGT) IU/L;
Biometric measure: Liver Function Test | At commencement (admission) to inpatient unit and after completion of follow up period at 3 months (12weeks)
  Outside of normal parameters (red flagged) Liver function test (LFTs) - components.
  • Aspartate aminotransferase (AST) IU/L;
Biometric measure: Liver Function Test | At commencement (admission) to inpatient unit and after completion of follow up period at 3 months (12weeks)
  Outside of normal parameters (red flagged) Liver function test (LFTs) - components.
  • Bilirubin mmol/L;
Biometric measure: Liver Function Test | At commencement (admission) to inpatient unit and after completion of follow up period at 3 months (12weeks)
  Outside of normal parameters (red flagged) Liver function test (LFTs) - components.
  • Total Protein Prothrombin Time (PT) g/L.
Biometric measures: Lipid Levels | At commencement (admission) to inpatient unit and after completion of follow up period at 3 months (12weeks)
  Outside of normal parameters (red flagged) Total Cholesterol ≥6.2mmol/L LDL (bad cholesterol) ≥4.1mmol/L HDL (good cholesterol) <2.1mmol/L Triglycerides ≥2.2mmol/L
Biometric measure: Glucose | At commencement (admission) to inpatient unit and after completion of follow up period at 3 months (12weeks)
  Outside of normal parameters (red flagged) <4.0 - >7.0 millimoles of glucose per litre of blood (mmols/L)
Biometric measure: Respiratory Rate | At commencement (admission) to inpatient unit and after completion of follow up period at 3 months (12weeks)
  Outside of normal parameters (red flagged) >20 Respiratory rate per minute (rpm)
Biometric measure: Sleep | At commencement (admission) to inpatient unit and after completion of follow up period at 3 months (12weeks)
  Outside of normal parameters (red flagged) Self reported: <3hours per night >8hours per night
Biometric measure: Smoking | At commencement (admission) to inpatient unit and after completion of follow up period at 3 months (12weeks)
  Outside of normal parameters (red flagged)
  Self reported:
  Smoker - volume per day Passive smoker Non-smoker
Biometric measure: Alcohol | At commencement (admission) to inpatient unit and after completion of follow up period at 3 months (12weeks)
  Outside of normal parameters (red flagged) Self reported: >units per day
Biometric measure: Fluid intake | At commencement (admission) to inpatient unit and after completion of follow up period at 3 months (12weeks)
  Outside of normal parameters (red flagged) Self reported: <1litre/day >3litres/day
Biometric measure: Caffeine intake | At commencement (admission) to inpatient unit and after completion of follow up period at 3 months (12weeks)
  Outside of normal parameters (red flagged) Self reported: ≥600milligrams (mg) /day
Biometric Measure: Urine output | At commencement (admission) to inpatient unit and after completion of follow up period at 3 months (12weeks)
  Outside of normal parameters (red flagged) Self reported: <1litre/day >2litres/day
Biometric measure: Bowel Function | At commencement (admission) to inpatient unit and after completion of follow up period at 3 months (12weeks)
  Outside of normal parameters (red flagged) Bristol Stool Scale
Biometric measure: Reproductive Health | At commencement (admission) to inpatient unit and after completion of follow up period at 3 months (12weeks)
  Outside of normal parameters (red flagged)
  Self reported:
  Sexual Transmitted Infection screening - recent/occasionally/never Female: menstrual cycle Regular 28day ovulation cycle (range:24---35 days) Male: prostate and testicular (self examination) recent/occasionally/never Sexual satisfaction: Satisfied/dissatisfied
Biometric measure: Diet | At commencement (admission) to inpatient unit and after completion of follow up period at 3 months (12weeks)
  Outside of normal parameters (red flagged) Intake (serving) per day of protein, fruit, vegetables
Biometric measure: Exercise | At commencement (admission) to inpatient unit and after completion of follow up period at 3 months (12weeks)
  Outside of normal parameters (red flagged) Self reported: minutes per day
Biometric measure: Eyes | At commencement (admission) to inpatient unit and after completion of follow up period at 3 months (12weeks)
  Outside of normal parameters (red flagged)
  Self reported:
  Concerns/no concerns
Biometric measure: Oral Health | At commencement (admission) to inpatient unit and after completion of follow up period at 3 months (12weeks)
  Outside of normal parameters (red flagged)
  Self reported:
  Concerns/no concerns

IPD SHARING:
Plan to Share IPD: No
Facility request not to share IPD

REFERENCES:
- [Background] Werkkala C, Valimaki M, Anttila M, Pekurinen V, Bressington D. Validation of the Finnish Health Improvement Profile (HIP) with patients with severe mental illness. BMC Psychiatry. 2020 Mar 11;20(1):112. doi: 10.1186/s12888-020-02511-5. PMID 32160873
- [Background] Meepring S, Gray R, Li X, Chien WT, Li Y, Ho GWK, Kritkitrat P, Bressington D. Evaluating the efficacy of the Thai Health Improvement Profile intervention for preventing weight gain in people with early stage psychosis: A randomized controlled trial. Int J Nurs Stud. 2023 Oct;146:104570. doi: 10.1016/j.ijnurstu.2023.104570. Epub 2023 Jul 31. PMID 37597457
- [Background] White J, Gray R, Jones M. The development of the serious mental illness physical Health Improvement Profile. J Psychiatr Ment Health Nurs. 2009 Jun;16(5):493-8. doi: 10.1111/j.1365-2850.2009.01375.x. Epub 2008 Mar 9. PMID 19538607